CLINICAL TRIAL: NCT03247777
Title: Benefits of Traditional and Golf-specific Resistance Training in Amateur Female Golfers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Point University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPU#201310-227
Record Dates: First submitted 2015-05-04; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Improved Performance in Amateur Female Golfers (MESH Term: Body Composition)
Keywords: golf; strength training; physical performance tests; body composition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional strengthening (Active Comparator): These subjects performed traditional strengthening exercises of targeted muscle groups (For example, bench press, lat pulldowns, dead lifts and wrist curls)
  Interventions: Other: Traditional strengthening
- Functional Strengthening (Active Comparator): These subjects performed exercises that either mimicked golf (diagonal chop) or that required balance and stability (single leg dead lift)
  Interventions: Other: Functional Strengthening

INTERVENTIONS:
Other: Traditional strengthening — dead lifts, bench press, wrist curls, and lat pulldowns as examples
  Arms: Traditional strengthening
Other: Functional Strengthening — diagonal chops, one leg deadlifts, lateral plyometrics as examples
  Arms: Functional Strengthening

SUMMARY:
Amateur female golfers were randomized to either a functional weight lifting group or a traditional weight lift group. Testing, consisting of performance measures and golf measures, was performed at baseline and after 10 weeks of weight lifting.

DETAILED DESCRIPTION:
A randomized control trial to compare the effects of 10 weeks of two different types of training in recreationally active female golfers was performed. Participants were recruited through postings at local country clubs and public golf courses, as well as through emails to state and local women's golf associations. Following written informed consent approved by the university's institutional review board, participants completed a medical and golf history questionnaire. Golf-specific information gathered via the history form included self-reported number of years playing golf, handicap, frequency of play, frequency of practice. Baseline testing followed, consisting of measurement of height and weight using a stadiometer, bone density and body composition using dual energy X-ray absorptiometry (DXA), 7-iron and driver club speed and total ball distance using a golf simulator (High Definition Golf, Interactive Sports Technologies, Vaughan, Ontario), and physical performance tests. Participants were then randomly assigned, using a random number generator, to either a traditional resistance training group (TRAD) or a golf-specific resistance training group (GSRT). Resistance training was conducted 3 days per week for 10 weeks. Each training session was directly supervised by at least one of the researchers, such that correct technique and appropriate resistance could be monitored. Following the 10 weeks of training, participants repeated the testing procedures under similar conditions as baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* females ≥18 years of age,
* and an official handicap or completion of at least 5 rounds of golf within the last year

Exclusion Criteria:

* Exclusion criteria were current episode of musculoskeletal pain,
* unable to stand and swing a golf club independently,
* systemic disease including but not limited to rheumatologic disease or cancer,
* or psychological or other cognitive impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Driver club speed | 10 weeks
  Driver club speed- continuous variable measured in mph
7-iron club speed | 10 weeks
  7-iron club speed-continuous variable measured in mph
Driver distance | 10 weeks
  Driver distance-continuous variable measured in yards
7-iron distance | 10 weeks
  7-iron -continuous variable measured in yards

SECONDARY OUTCOMES:
Seated rotation flexibility | 10 weeks
  sit and rotate left and right- continuous variable measured with a goniometer in degrees
Weighted ball golf toss | 10 weeks
  Using a golf-like motion, toss a 6lb ball as far as possible- continuous scale measured in cm
Weighted ball seated toss | 10 weeks
  sitting in a declined position, use a chest pass motion to toss a 6 lb ball as far as possible- continuous measure measured in cm

OTHER OUTCOMES:
Bone density | 10 weeks
  bone density- continuous measure measured using a dual image x-ray absorptiometry (DEXA) scan
Body fat percentage | 10 weeks
  body fat percentage- 0-100% scale measured using a DEXA scan

CONTACTS AND LOCATIONS:
Locations (1):
- Human Biomechanics and Physiology Study, High Point, North Carolina, United States